CLINICAL TRIAL: NCT01691404
Title: Study on the Effects of Epicatechin and Quercetin Supplementation on Vascular Function and Blood Pressure in Untreated (Pre)Hypertensive Subjects
Brief Title: Study on the Effects of Epicatechin and Quercetin Supplementation on Vascular Function and Blood Pressure (FLAVO)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: Top Institute Food and Nutrition (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: NL4077208112
Record Dates: First submitted 2012-09-12; First posted 2012-09-24 (Estimated); Last update posted 2013-04-23 (Estimated); Status verified 2012-11

CONDITIONS: Hypertension; Endothelial Dysfunction
Keywords: Flavonoids; Quercetin; Epicatechin; Vascular function; Blood pressure; Endothelial function
MeSH Terms: conditions — Hypertension | interventions — Catechin; Quercetin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Epicatechin (Active Comparator): Subjects will be asked to consume supplements containing 100mg of epicatechin daily
  Interventions: Dietary Supplement: Epicatechin
- Quercetin (Active Comparator): Subjects will be asked to consume supplements containing 160mg of quercetin-3-glucoside daily
  Interventions: Dietary Supplement: Quercetin
- Placebo (Placebo Comparator): Subjects will be asked to consume capsules containing a placebo (cellulose) daily
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Epicatechin — Subjects will be asked to consume supplements containing 100mg of epicatechin daily
  Arms: Epicatechin
Dietary Supplement: Quercetin — Subjects will be asked to consume 160mg of quercetin-3-glucoside daily
  Arms: Quercetin
Dietary Supplement: Placebo — Subjects will be asked to consume capsules containing placebo (cellulose) daily
  Arms: Placebo

SUMMARY:
Flavonoid-rich foods such as tea and cocoa have been identified as having a blood pressure-lowering effect. Part of this effect is thought to be due to the flavonoid content of these foods although it is currently unknown which flavonoids play a role. Epicatechin is one the major flavonoids in cocoa while quercetin is largely found in tea.

During this study the investigators plan to investigate the effects of pure epicatechin and quercetin supplementation on vascular function and blood pressure in untreated (prehypertensive) subjects by way of a three-armed double-blind crossover intervention. Participants will sequentially consume supplements containing quercetin, epicatechin or placebo for a period of 4 weeks. Before and after this 4 week period, measurements of vascular function and blood pressure will be taken.

The investigators hypothesize that the supplementation of epicatechin and quercetin will improve vascular function and blood pressure.

DETAILED DESCRIPTION:
By means of a three-armed double-blind crossover intervention, the effects of pure flavonoid supplementation will be investigated. The products under investigation will be epicatechin and quercetin-3-glucoside. Subjects will be asked to consume either 160mg of quercetin-3-glucoside, 100mg of epicatechin or a placebo capsule for a period of 4 weeks. Measurements of vascular function and blood pressure will be taken before and after each 4-week intervention period. A 4-week washout period will be planned between each intervention.

Measurements of vascular function will include flow-mediated dilation, pulse wave analysis, pulse wave velocity and vasomotion as well as biomarkers of inflammation and vascular function.

ELIGIBILITY:
Inclusion Criteria:

* Systolic Blood Pressure between 125 and 160 mmHg
* Age between 30 and 80 years
* BMI > 20 and ≤ 40
* No reported current or previous metabolic diseases
* No history of cardiovascular diseases
* No history of renal, liver or thyroid diseases
* No history of gastrointestinal diseases
* No diabetes mellitus
* Fasting laboratory parameters within normal range: complete blood count (RBC, WBC, PLT, HB, HT), renal function (serum creatinine, urea), liver function (ALAT, ASAT, ɣ-GT), and serum glucose.

Exclusion Criteria:

* Body mass index > 40 and ≤20
* Secondary hypertension
* Weight loss or weight gain of 5 kg or more during the last 2 months
* Usage of non-steroidal anti-inflammatory drugs (acetylsalicylic acid, ibuprofen, naproxen) and not able or willing to stop taking them from at least 4 weeks prior to the study
* Usage of cholesterol-lowering medication
* Daily usage of corticosteroids
* Medical treatment that may affect blood pressure and not able (or willing) to stop
* Taking nutritional supplements and unwilling to discontinue
* Lactating, pregnant or intention to become pregnant during study
* Reported dietary habits, medically prescribed diet, slimming diet
* Reported average alcohol consumption > 2 glasses/d (men) or >1 glass/d (women)
* Problems with consuming the supplements or following the study guidelines
* Unwilling to undergo home or office blood pressure measurements
* Recent blood donation i.e. 1 month (male subjects) or 2 months (female subjects) prior to the study and planned donation during the study period
* Reported intense sporting activities > 10 h/w
* Not agreeing to be informed about unexpected and medically relevant personal test-results, or not agreeing that their general practitioner will be informed about these results
* Participation in another biomedical trial less than 2 months before the start of the study or at the same time
* No signed informed consent form
* Clinical disorders that could interfere with the intervention
* Unable to comply with the study procedure (e.g. holidays, urine collection, blood sampling)
* Smokers
* Difficulty imaging brachial artery by ultrasonography

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2012-09; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Change in Endothelium-dependent flow-mediated dilation as a result of epicatechin and quercetin-3-glucoside supplementation | Baseline and every 4 weeks thereafter (weeks 4, 8, 12, 16 and 20)
  Change in arterial diameter as a result of 5 minute arterial occlusion (200mmHg). Arterial diameter will be measured by means of ultrasonography.

SECONDARY OUTCOMES:
Change in blood pressure as a result of epicatechin and quercetin-3-glucoside supplementation | Baseline and every 4 weeks thereafter (weeks 4, 8, 12, 16 and 20)
  Office BP (Dinamap, 4 consecutive measurements with 2-min intervals)and 24-hour ABPM (Spacelab; 1x24h)
Change in pulse wave velocity as a result of epicatechin and quercetin supplementation | Baseline and every 4 weeks thereafter (weeks 4, 8, 12, 16 and 20)
  Measured using a SphygmoCor device at baseline and the end of each intervention
Change in vasomotion as a result of epicatechin and quercetin supplementation | Baseline and every 4 weeks thereafter (weeks 4, 8, 12, 16 and 20)
  Measured using a PeriFlux 5001 device at baseline and the end of each intervention.
Changes in biomarkers of endothelial function as a result of epicatechin and quercetin supplementation | Baseline and every 4 weeks thereafter (weeks 4, 8, 12, 16 and 20)
  Plasma analysis of endothelin-1, ADMA, MCP-1, sVCAM-1, sICAM-1, sE-selectin, sTM, CRP, SAA, IL-6, IL-8, TNF-α, vWF, nitric oxide
Changes in peripheral blood mononuclear cell gene expression of markers of inflammation as a result of epicatechin and quercetin supplementation | Baseline and every 4 weeks thereafter (weeks 4, 8, 12, 16 and 20)
  PBMC gene expression of markers of inflammation
Change in cardiovascular parameters in plasma as a result of epicatechin and quercetin supplementation | Baseline and every 4 weeks thereafter (weeks 4, 8, 12, 16 and 20)
  Total cholesterol, HDL-cholesterol, LDL-cholesterol, triglycerides, insulin and glucose
Changes in pulse wave analysis as a result of epicatechin and quercetin supplementation | Baseline and every 4 weeks thereafter (weeks 4, 8, 12, 16 and 20)
  Measured using a SphygmoCor device at baseline and the end of each intervention
Adverse events | Baseline and every 2 weeks thereafter (weeks 2, 4, 6, 8, 10, 12, 14, 16, 18 and 20)
  During the study subjects will be asked to maintain a diary in which they can report any adverse events they may have a result of the supplements. Diaries will be checked every 2 weeks. Study subjects will also be asked to contact the research team if they experience repeated adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hollman, PhD, Principal Investigator — Wageningen University
Locations (1):
- Wageningen University, Wageningen, Netherlands

REFERENCES:
- [Derived] Van den Eynde MDG, Geleijnse JM, Scheijen JLJM, Hanssen NMJ, Dower JI, Afman LA, Stehouwer CDA, Hollman PCH, Schalkwijk CG. Quercetin, but Not Epicatechin, Decreases Plasma Concentrations of Methylglyoxal in Adults in a Randomized, Double-Blind, Placebo-Controlled, Crossover Trial with Pure Flavonoids. J Nutr. 2018 Dec 1;148(12):1911-1916. doi: 10.1093/jn/nxy236. PMID 30398646
- [Derived] Dower JI, Geleijnse JM, Gijsbers L, Schalkwijk C, Kromhout D, Hollman PC. Supplementation of the Pure Flavonoids Epicatechin and Quercetin Affects Some Biomarkers of Endothelial Dysfunction and Inflammation in (Pre)Hypertensive Adults: A Randomized Double-Blind, Placebo-Controlled, Crossover Trial. J Nutr. 2015 Jul;145(7):1459-63. doi: 10.3945/jn.115.211888. Epub 2015 May 13. PMID 25972527
- [Derived] Dower JI, Geleijnse JM, Gijsbers L, Zock PL, Kromhout D, Hollman PC. Effects of the pure flavonoids epicatechin and quercetin on vascular function and cardiometabolic health: a randomized, double-blind, placebo-controlled, crossover trial. Am J Clin Nutr. 2015 May;101(5):914-21. doi: 10.3945/ajcn.114.098590. Epub 2015 Feb 25. PMID 25934864
- See also: Website for the study (in dutch) — http://voedingsonderzoek.wur.nl/flavo